CLINICAL TRIAL: NCT00345462
Title: Immunogenicity and Reactogenicity of Trivalent Virosomal Influenza Vaccine Invivac® for the Season 2006/2007. An Open, Baseline-controlled Study in Two Groups of Healthy Subjects: Adults and Elderly.
Brief Title: Annual Study to Investigate Inactivated Virosomal Influenza Vaccine for the 2006/2007 Influenza Season in Europe.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S206.3.012; 2006-001301-28
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Healthy Volunteers
Keywords: Influenza, Vaccine, CHMP criteria
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Trivalent virosomal influenza vaccine

SUMMARY:
Influenza (flu) viruses change continuously, therefore also the parts of viruses used in influenza vaccines can vary from year to year. In Europe, manufacturers/marketing holders of these vaccines are required to be involved in ongoing clinical trials and to present the results to the competent authorities each year. The current study is a phase IIIa clinical trial with a commercially available virosomal vaccine (Invivac®) supplied in pre filled syringes. It is part of the ongoing clinical trial program for Invivac® and will be done to assess the immunogenicity and safety and tolerability of next season's trivalent influenza virosomal vaccine in two groups of healthy subjects: subjects aged >= 18 and <= 60 years and subjects >= 61 years of age (elderly).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent.
* Healthy and aged >= 18 and <= 60 years or >= 61 years of age.
* Mental health good enough to understand the study and the informed consent form and to fill in the questionnaire."

Exclusion Criteria:

* Known to be allergic to eggs, chicken protein, gentamicin or any other constituent of the vaccine.
* Having fever and/or presenting with an acute infectious episode of the upper and/or lower respiratory airways.
* Having experienced a documented serious systemic reaction after previous influenza vaccination.
* Having an auto-immune disorder (e.g. RA, SLE, auto-immune thyroid disorders) or other disorders affecting the immune system, taking immunosuppressive medication (such as systemic corticosteroids) including the four weeks preceding the start of the study (date of informed consent), or having a disease in a terminal stage.
* Having received vaccination against influenza within the previous six months before Visit 1.

Exclusion criteria only for female subjects aged >=18 and <=60 years and of childbearing potential:

* Pregnancy (positive urine pregnancy test on Day 1) or breastfeeding.
* Absence of use of a medically accepted method of birth control (i.e. oral contraceptive, Intra Uterine Device, double barrier method).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-06

PRIMARY OUTCOMES:
Immunogenicity (HI-titers after 2 and 3 weeks), reactogenicity and inconvenience of Invivac® 2006/2007

SECONDARY OUTCOMES:
HI derived parameters: seroprotection, seroconversion and mean fold increase (CHMP)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, Berlin, Germany